CLINICAL TRIAL: NCT05102981
Title: StomaFUNQ. Function and Quality of Life After Emergency vs Planned Creation of a Stoma
Brief Title: Function and Quality of Life After Emergency vs Planned Creation of a Stoma
Acronym: StomaFUNQ
Status: Enrolling by invitation | Type: Observational
Sponsor: Eva Haglind, MD, PhD, professor (Other)
Responsible Party: Sponsor-Investigator, Eva Haglind, MD, PhD, professor, Professor emerita, Consultant, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Other Study IDs: 2021-04078
Record Dates: First submitted 2021-10-18; First posted 2021-11-02 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- emergency stoma: an emergency procedure including stoma construction, as first procedure at or shortly after diagnosis of colon or rectal cancer
  Interventions: Procedure: emergency procedure
- Planned stoma: a planned procedure including stoma construction, as first procedure after diagnosis of colon or rectal cancer
  Interventions: Procedure: emergency procedure

INTERVENTIONS:
Procedure: emergency procedure — The difference between groups is the timing or type ie emergency as opposed to planned

SUMMARY:
The aim is to compare functional outcome and or quality of life in patients with a stoma that was constructed as an emergency procedure with patients where a stoma was created as a planned procedure. To do this data will be retrieved from the Swedish Patient Register to identify all patients with a diagnosis of colorectal cancer and a stoma construction procedure during two previous calender years. To collect data on stoma function and quality of life a specific questionnaire will be sent to the cohort approximately within 2 years of the procedure.

DETAILED DESCRIPTION:
The cohort will be identified through the National in-Patient Register, held by the Swedish Board of Health and Welfare, by using a combination of ICD10 and NOMESCO codes. Two calender years will be the collecytion period to reach group size allowing for statistical analysis. Data from the register will be used to describe the groups (demography) and data from the prescribed drug register to calculate costs for stoma appliances after discharge.

Using the patient ID, all patients still alive at the time, will be contacted first by a letter followed within 2-4 days by a phomecall from the study secretariate, to ask for consent and thereafter to send out the questionnaire.

The questionnaire includes validated questions used before as well as validated instruments, to analyze stoma function in detail as well as quality fo life, as well as questions where answers will be used for adjustment in analyses.

ELIGIBILITY:
Inclusion Criteria:

* stoma permanently or for shorter period

Exclusion Criteria:

* not understanding Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all registered individuals who had a primary surgical procedure including a stoma as treatemtn for colon or rectal cancer in Sweden in 2019 and 2020.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Function of stoma | < 3 years of creation
  rate of patients who are satisfied with stoma function
function of stoma | <3 years of stoma creation
  rate of patients experiencing leakage from stoma appliance

SECONDARY OUTCOMES:
Patient reported quality of life | 3 years after of stoma creation
  Patient reported quality of life by question: "How was your quality of life during the last month?" answered through a 7 step Likert scale anchored by "worst possible" and "best possible"

OTHER OUTCOMES:
cost of stoma care | < 3 years of stoma construction
  health economic analysis of costs such as of stoma appliances, visits to stoma nurses, re-operations to improve stoma and/or repair a parastomal hernia

CONTACTS AND LOCATIONS:
Locations (1):
- Gothenburg University, Sahlgrenska Academy, Institute of Cinical Sciences, Department of Surgery, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No